CLINICAL TRIAL: NCT03210090
Title: Impact of the Lack of CMV-Specific CD8+ T Cell Response in CMV-Seropositive Donors in CMV Reactivation After Hematopoietic Stem Cells Transplant in CMV-Seropositive Recipients
Acronym: CYTHEMAT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Maimónides Biomedical Research Institute of Córdoba (Other)
Collaborators: QIAGEN Gaithersburg, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: HSCT-CMV-2015-01
Record Dates: First submitted 2017-04-25; First posted 2017-07-06 (Actual); Last update posted 2017-07-06 (Actual); Status verified 2017-07

CONDITIONS: Cytomegalovirus Infection; HSCT
Keywords: Stem cells transplantation; Cytomegalovirus infection; CMV-Specific Immune response; Immune reconstitution; Humoral/Cellular mismatch; Interferon-gamma
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Donor and recipient CMV-serostatus is one of the risk factor for CMV infection in solid organ transplantation. Recipients with IgG positive anti-CMV are classified as low-risk patients since it is considered that patients also have specific cellular immunity against CMV. However, investigators group has published that around 25% of solid organ transplant candidates lack CMV-specific CD8+ T-cell response ("humoral/cellular mismatch") and they are at a higher risk of CMV replication after transplantation. The main goal of this study is to analyze the impact of the humoral/cellular mismatch in hematopoietic stem cell transplantation (HSCT) CMV-seropositive donors on the CMV reactivation after HSCT in CMVseropositive recipients. Investigators will study not only the incidence of CMV reactivation but also the severity (duration and peak viral load), CMV disease and survival. CMV-seropositive patients who receive a HSCT (bone marrow or peripheral blood) from related donors will be consecutively recruited from Reina Sofía Hospital (Córdoba) and Marqués de Valdecilla Hospital (Santander).

Patients will be monitored during 12 months after HSCT. CMV-specific CD8+ T-cell response will be determined in their donors, using QuantiFERON-CMV assay, to know the frequency of humoral/cellular mismatch. Innate and adaptive immune reconstitution will be assessed by flow cytometry and experimental QuantiFERON Monitor assay. CMV-specific CD8+ T-cell reconstitution will be determined using QuantiFERON-CMV assay.

ELIGIBILITY:
Inclusion Criteria:

1. CMV Seropositive patients who receive a HSCT (Bone marrow or peripheral) blood from related donors
2. >14 years old
3. signed Inform consent form

Exclusion Criteria:

1. HIV, HCV, HBV Infection

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: CMV-seropositive patients who receive a HSCT (bone marrow or peripheral blood) from related donors.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2016-01-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
To determine the incidence and severity of CMV reactivation in CMV-seropositive patients whose stem cells come from CMV seropositive donors lacking CMV-specific CD8+ T-Cell response [D+(T-)/R+] in comparison with D+(T+)/R+ and D-/R+ patients | During the 6 months after transplantation
  To determine the incidence and severity of CMV reactivation in CMV-seropositive patients whose stem cells come from CMV seropositive donors lacking CMV-specific CD8+ T-Cell response [D+(T-)/R+] in comparison with D+(T+)/R+ and D-/R+ patients

SECONDARY OUTCOMES:
To analyze the frequency of CMV-seropositive stem cells donors lacking CMV-specific CD8+ T-Cell response [D+(T-)] | 3 years
  To analyze the frequency of CMV-seropositive stem cells donors lacking CMV-specific CD8+ T-Cell response [D+(T-)]
Innate and adaptive immune reconstitution: Units (percentage and absolute number) | 3 years
  To analyze the differences in the innate, adaptive as well as CMV-specific immune reconstitution between D+(T-)/R+ vs D-/R+ and D+(T+)/R+ patients
To evaluate the incidence of CMV disease as well as the type and severity of the disease in D+(T-)/R+ vs D-/R+ and D+(T+)/R+ patients | 3 years
  To evaluate the incidence of CMV disease as well as the type and severity of the disease in D+(T-)/R+ vs D-/R+ and D+(T+)/R+ patients
CMV-specific immune reconstitution: Units (Percentage respect to CD8+ T cells) and interferon-gamma production (IU/mL). | 3 years
  To test the differences in mortality/survival between the three groups

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Hospital Marques de Valdecilla, Santander, Cantabria
  - Hosìtal Universitario Reina Sofia, Córdoba

IPD SHARING:
Plan to Share IPD: No